CLINICAL TRIAL: NCT01465191
Title: Effect of OPRM1 Genotype on the Dose Response to Spinal Morphine for Post-Cesarean Analgesia
Brief Title: Effect of Mu-opioid Receptor Genetics on 3 Doses of Spinal Morphine for Postoperative Analgesia After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Richard M. Smiley, Professr of Clinical Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAI2804
Record Dates: First submitted 2011-11-02; First posted 2011-11-04 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain
Keywords: cesarean; postoperative; morphine; genetics; opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 micrograms (mcg) spinal morphine (Experimental): Subjects will receive 50 mcg morphine in their spinal anesthetic for cesarean section
  Interventions: Drug: Morphine
- 100 micrograms spinal morphine (Experimental): Subjects will receive 100 mcg morphine in their spinal anesthetic for cesarean section
  Interventions: Drug: Morphine
- 150 micrograms spinal morphine (Experimental): Subjects will receive 150 mcg morphine in their spinal anesthetic for cesarean section
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section

SUMMARY:
HYPOTHESIS: The response to a given dose of morphine given via a spinal anesthetic for cesarean section will be affected by the genetics of the woman's mu-opioid receptor

Most women undergoing elective cesarean section (CS) receive spinal anesthesia, and most receive a dose of preservative free morphine with the spinal anesthetic. Spinally-administered morphine provides 16-24 hours of high quality pain relief. The dose administered is usually 75-200 micrograms, but surprisingly few dose-response studies exist.

The mu-opioid receptor (OPRM1 gene)is the site of action of endogenous opioid peptides and opioid analgesic drugs like morphine. There is a common genetic variant of this receptor at the 40th amino acid of the protein, with asparagine and asparate being present in different people. The less common variant (aspartate), present in 25-30% of the overall American population (higher in Asian populations, lower in Blacks) at codon 40 that has been shown in many studies to affect opioid analgesia.

This will be a randomized, blinded study of 3 doses of spinal morphine (50, 100, 150 micrograms) given to women undergoing elective cesarean section at term pregnancy. 300 women will be studied (100 per dose). Blood will be obtained for genotyping of OPRM1 and other genes that may affect pain and analgesic responses. The primary outcome will be the amount of intravenous morphine patients self-administer in the 24 hours postsurgery.

The primary outcome (use of intravenous morphine) will be analyzed by dose, and within each dose group by genotype of OPRM1. Secondary outcomes will include pain scores every 6 hours, satisfaction with analgesia, side effects (itching, nausea/vomiting) by dose and genotype.

It is anticipated that there will be an interim data analysis at 150 evaluable subjects for assessment of the dose response to morphine in the overall population; then a final analysis at 300 subjects for the genetic effect assessment.

ELIGIBILITY:
Inclusion Criteria:

* healthy women undergoing elective cesarean

Exclusion Criteria:

* cardiovascular disease
* analgesic medications
* complications of pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Smiley, MD, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 Micrograms Spinal Morphine: Subjects will receive 50 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed.
- 100 mcg Spinal Morphine: Subjects will receive 100 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed.
- 150 mcg Spinal Morphine: Subjects will receive 150 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed.
Period: Overall Study
Arm/Group | 50 Micrograms Spinal Morphine | 100 mcg Spinal Morphine | 150 mcg Spinal Morphine
Started | 56 | 63 | 50
Completed | 47 | 54 | 43
Not Completed | 9 | 9 | 7
Not completed — Protocol Violation | 6 | 3 | 3
Not completed — Lost to Follow-up | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- 50 Micrograms Spinal Morphine: these subjects will receive 50 mcg spinal morphine
- 100 Micrograms Spinal Morphine: these subjects will receive 100 mcg spinal morphine
- 150 Micrograms Spinal Morphine: these subjects will receive 150 mcg spinal morphine
- Total: Total of all reporting groups
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine | Total
Number analyzed (Participants) | 47 | 54 | 43 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 54 | 43 | 144
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6) | 33 (5) | 33 (6) | 33 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 54 | 43 | 144
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 54 | 43 | 144

OUTCOME MEASURES:

1. Primary Outcome: Milligrams of Intravenous Morphine Used by Participant in First 24 Hours Postoperatively
Description: IV morphine use in milligrams, by participant-controlled analgesia will be assessed every 6 hours for 24 hours postoperatively.
Time Frame: 24 hours
Measure: Mean (Inter-Quartile Range); unit: Milligrams
Groups:
- 50 Micrograms Spinal Morphine: Subjects will receive 50 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
Milligrams | 18 [8 to 29] | 14 [6 to 27] | 15 [5 to 23]

2. Secondary Outcome: Visual Analog Scale (VAS) Pain at 6 Hours
Description: Visual analog pain scale measures pain on a 100 millimeter (mm) scale. Participants make a mark on the scale with one end labeled "None" (0mm) and the other labeled "Worst pain imaginable" (100mm). Pain measured at rest and with movement.
Time Frame: 6 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Groups:
- 100 Micrograms Spinal Morphine: Subjects will receive 100 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed.
- 150 Micrograms Spinal Morphine: Subjects will receive 150 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed.
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm
  Rest | 20 [10 to 39] | 25 [8 to 43] | 15 [2 to 35]
  Movement | 43 [27 to 62] | 43 [28 to 65] | 30 [13 to 52]

3. Secondary Outcome: Visual Analog Scale (VAS) Pain at 12 Hours
Description: as for outcome 2
Time Frame: 12 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm
  Rest | 20 [0 to 35] | 15 [0 to 36] | 10 [3 to 22]
  Movement | 30 [10 to 60] | 35 [17 to 63] | 30 [11 to 62]

4. Secondary Outcome: Visual Analog Scale (VAS) Pain at 18 Hours
Description: as for outcome 2
Time Frame: 18 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm
  Rest | 17 [0 to 35] | 11 [0 to 28] | 5 [0 to 19]
  Movement | 32 [10 to 50] | 30 [0 to 40] | 26 [0 to 40]

5. Secondary Outcome: Visual Analog Scale (VAS) Pain at 24 Hours
Description: as for outcome 2
Time Frame: 24 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm
  Rest | 24 [9 to 43] | 21 [6 to 50] | 18 [0 to 32]
  Movement | 43 [22 to 65] | 41 [21 to 68] | 41 [21 to 68]

6. Secondary Outcome: Visual Analog Scale- Nausea/Vomiting at 6 Hours
Description: Visual analog nausea/vomiting scale measures nausea and vomiting on a 100mm scale. Participants make a mark on the scale with one end labeled "None" (0mm) and the other labeled "Worst Nausea/Vomiting Imaginable" (100mm).
Time Frame: 6 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 0 [0 to 15] | 7 [0 to 40] | 0 [0 to 40]

7. Secondary Outcome: Visual Analog Scale- Nausea/Vomiting at 12 Hours
Description: as for outcome 6
Time Frame: 12 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 0 [0 to 5] | 0 [0 to 6] | 0 [0 to 10]

8. Secondary Outcome: Visual Analog Scale- Nausea/Vomiting at 18 Hours
Description: as for outcome 6
Time Frame: 18 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 0 [0 to 2] | 0 [0 to 0] | 0 [0 to 0]

9. Secondary Outcome: Visual Analog Scale- Nausea/Vomiting at 24 Hours
Description: as for outcome 6
Time Frame: 24 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 0]

10. Secondary Outcome: Visual Analog Scale Pruritus (Itching) at 6 Hours
Description: Visual analog pruritus scale measures itching on a 100mm scale. Participants make a mark on the scale with one end labeled "None" (0mm) and the other labeled "Worst Itching Imaginable" (100mm).
Time Frame: 6 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 21 [10 to 45] | 37 [3 to 73] | 39 [19 to 65]

11. Secondary Outcome: Visual Analog Scale Pruritus (Itching) at 12 Hours
Description: as for outcome 10
Time Frame: 12 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 10 [0 to 20] | 23 [0 to 64] | 25 [0 to 45]

12. Secondary Outcome: Visual Analog Scale Pruritus (Itching) at 18 Hours
Description: as for outcome 10
Time Frame: 18 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 9 [0 to 20] | 13 [0 to 47] | 5 [0 to 25]

13. Secondary Outcome: Visual Analog Scale Pruritus (Itching) at 24 Hours
Description: as for outcome 10
Time Frame: 24 hours post-operatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 7 [0 to 16] | 12 [0 to 39] | 6 [0 to 30]

14. Secondary Outcome: Visual Analog Patient Satisfaction With Analgesia at 24 Hours
Description: Visual analog patient satisfaction scale measures satisfaction with analgesia on a 100mm scale. Participants make a mark on the scale with one end labeled "Completely Dissatisfied" (0mm) and the other labeled "Completely Satisfied" (100mm).
Time Frame: 24 hours postoperatively
Measure: Mean (Inter-Quartile Range); unit: mm
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
Number analyzed (Participants) | 47 | 54 | 43
mm | 85 [65 to 100] | 83 [67 to 100] | 84 [70 to 100]

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- 50 Micrograms Spinal Morphine: Subjects will receive 50 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed and analyzed with 47 in this group
- 100 Micrograms Spinal Morphine: Subjects will receive 100 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed and analyzed with 54 in this group
- 150 Micrograms Spinal Morphine: Subjects will receive 150 mcg morphine in their spinal anesthetic for cesarean section
  Morphine: Morphine will be given via spinal injection at doses of 50, 100, 150 micrograms as part of a spinal anesthetic for cesarean section
  After interim analysis, the genetics part of the analysis was dropped and the study completed and analyzed with 43 in this group
Arm/Group | 50 Micrograms Spinal Morphine | 100 Micrograms Spinal Morphine | 150 Micrograms Spinal Morphine
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/54 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/54 | 0/43
Other Adverse Events (participants affected / at risk) | 0/47 | 0/54 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No